CLINICAL TRIAL: NCT00652600
Title: Comparative, Randomized, Single-Dose, 2 Way Cross Over Bioavailability Study of Par Propranolol 160 mg With That of Inderal-LA Propranolol 160 mg in Healthy Subjects Under Fed Conditions.
Brief Title: Bioavailability Study of Propranolol Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: SFBC Anapharm (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 50233
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: Bioequivalence, Propranolol ER capsules, fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Par formulated product under fed conditions
  Interventions: Drug: Propranolol
- B (Active Comparator): Subjects received Wyeth Pharmaceuticals formulated product under fed conditions
  Interventions: Drug: Inderal-LA

INTERVENTIONS:
Drug: Propranolol — ER Capsules, 160 mg, single-dose
  Other Names: Inderal-LA
  Arms: A
Drug: Inderal-LA — ER Capsules, 160 mg, single-dose
  Other Names: Propranolol ER capsules
  Arms: B

SUMMARY:
To compare the single-dose bioavailability of Propranolol 160 Mg ER Capsules with Inderal-La

DETAILED DESCRIPTION:
To compare the single -dose bioavailability of Par Propranolol 160 Mg ER capsules with Wyeth Pharmaceuticals, Inderal-LA, Propranolol under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the study will be members of the community at large. The Recruitment advertisements may use various media types (E.g. ratio, newspapers, SFBC Anapharm Website, SFBC Anapharm volunteer's database). Subjects must meet all the following criteria in order to be included in the study.
* Male and female, non-smoker, 18 years of age and older
* Capable of consent
* BMI ≥ 19.0 and > 30.0 kg/ m2.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study.
* Clinically significant illness within 4 weeks prior to the administration of the study medication
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub- Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or heart rate less than 60 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [ 1 Unit = 150mL of wine, 360 mL of beer, or 45mL of 40% alcohol])
* Use of soft drugs ( such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug at screening.
* History of allergic reactions to heparin, propranolol, or other related drugs.

  --Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin,glucocorticoids, omerprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known as interface with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of a study medication or over the counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptive.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 6 months proceeding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub- Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than contraceptives) within 3 months prior to administration of study medication.
* Donation of plasma (500 Ml) within 7 days to drug administration. Donation or loss of hole blood (excluding the volume of blood drawn during the screening procedures of this study) prior to administration of the study medication as follows.
* 50mL to 300mL of whole blood within 30 days, 301 mL to 500 ml of whole blood within 45days or more than 500 mL of whole blood within 56 days prior to drug administration..
* History bronchial asthma and bronchospastic diseases.
* History of known presence of cardiogenic shock, sinus bradycardia, Wolff-Parkinson White Syndrome, congestive heart failure or angina.
* Clinically significant history of diabetes.
* Clinically significant history of hyperthyroidism.
* Breast- feeding subject.
* Positive urine pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non- sterile male partner (i.e. male who ahs not been sterilized by vasectomy for al least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception:
* Intra-uterine contraceptive device (place al least 4 weeks prior to study drug administration)
* Condom or diaphragm. + spermicide
* Hormonal contraceptives (starting al least 4 weeks prior to study administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, Principal Investigator — SFBC Anapharm